CLINICAL TRIAL: NCT04520139
Title: Phase I Dose-Escalating and Phase II Dose-Expansion Study of N-Acetyl-Cysteine (NAC) Administration to Ovarian Cancer Patients Receiving Platinum-Based Therapy (PBT) for the Mitigation of Chemotherapy-Related Cognitive Impairment (CRCI)
Brief Title: Effect of NAC on Preventing Chemo-Related Cognitive Impairments in Ovarian Ca Pts Treated W/ PBT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Jarrow Formulas Inc (Industry)
Responsible Party: Principal Investigator, Daniela A. Bota, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20205846; UCI 18-120 (Other: Chao Family Comprehensive Cancer Center)
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Cognitive Impairment
Keywords: Chemotherapy-Related Cognitive Impairments
MeSH Terms: conditions — Ovarian Neoplasms; Cognitive Dysfunction; Chemotherapy-Related Cognitive Impairment | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Phase 1 will be a dose-escalating design.
  Phase 2 will be a randomized, double-blinded, placebo-controlled study design
Who Masked: Participant, Investigator
Masking Description: Phase 1 will be open label.
  Phase 2 will be be double-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Patients will receive NAC beginning at Cohort 1. If, at a given dose, none of the 3 patients shows a dose-limiting toxicity during the first cycle of PBT, then the dose is escalated 1 step for subsequent subjects. If, at a given dose, only 1 of 3 shows a dose-limiting toxicity, then up to 3 additional participants will be enrolled at that dose.If, at a given dose, the first 2, or any 2 of 3 subjects show a dose-limiting toxicity, then the dose will be de-escalated 1 step for future participants. At a dose where enrollment is expanded to between 4 and 6, if only 1 of 6 subjects shows a dose-limiting toxicity, then the dose will be escalated 1 step for future participants. However, if 2 or more of 4, 5, or 6participants show a dose-limiting toxicity, then the dose will be reduced one step for future participants. The maximum tolerated dose is defined as the highest dose not requiring deescalation. This is the dose to be used for the NAC arm of Phase II study.
  Interventions: Drug: N-Acetyl-Cysteine
- Phase 2 Dose Expansion (Experimental): Patients will be randomized to receive NAC at the maximum tolerated dose or placebo.
  Interventions: Drug: N-Acetyl-Cysteine; Other: Placebo

INTERVENTIONS:
Drug: N-Acetyl-Cysteine — Given PO
  Other Names: NAC Sustain; NAC
Other: Placebo — Given PO
  Arms: Phase 2 Dose Expansion

SUMMARY:
This is a phase I, dose-escalation and phase II dose-expansion clinical trial determining the maximum tolerated dose (MTD) and safety and tolerability of adding N-Acetyl-Cysteine (NAC) to ovarian cancer patients who are receiving a platinum-based therapy (PBT). This study will investigate whether NAC will mitigate chemotherapy-related cognitive impairment (CRCI).

ELIGIBILITY:
Inclusion Criteria:

Post-menopausal females (as defined by lack of menstruation for 12 months or status post oophorectomy)

* Histologic or pathologic diagnosis of stage III-IV epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Eastern Cooperative Oncology Group (ECOG) ≤2
* Life expectancy > 1 year
* Status post cytoreductive surgery for ovarian cancer or with planned cytoreductive surgery if treated with neoadjuvant chemotherapy
* Prescribed a minimum of six cycles of platinum-based chemotherapy
* Adequate organ function as defined below:

  1. Hemoglobin > 9 g/dL
  2. Leukocytes >1,500/mcl
  3. Absolute Neutrophil Count > 1,000/mcL
  4. Platelets > 125,00/mcL
  5. total bilirubin Within normal institutional limits
  6. Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 x institutional upper limit of normal
  7. Serum creatinine < 1.5 mg/dL.

Exclusion Criteria:

* Prior history of any cancer (other than non-melanoma skin cancer)
* Chemotherapy, radiation therapy, or erythropoietin treatment within the last 6 months
* Prior severe head injury
* Has a history of dementia or other neurodegenerative disorders
* Has an uncontrolled, treatment-resistant depression or other severe psychiatric illnesses
* Presence of known brain metastases
* Has an active infection requiring treatment
* Known immunosuppressive disease
* Has active systemic autoimmune diseases such as lupus
* Receipt of systemic immunosuppressive therapy
* Known human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C
* Pregnant of breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study targets post-menopausal women with a histologically confirmed diagnosis of stage III-IV eipithelial ovarian cancer, fallopian tube, or primary peritoneal cancer
Enrollment: 102 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of N-Acetyl-Cysteine in Ovarian Cancer Patients Receiving Platinum-Based Therapy | From the start date of treatment until 6 months after removal of treatment due to toxicity, termination of study or withdrawal of treatment, whichever came first.
  Determination of the maximum tolerated dose (MTD) will be utilized to evaluate the safety and tolerability of adding N-Acetyl-Cysteine (NAC) in ovarian cancer patients who are also receiving platinum-based therapy (PBT), using a Phase I, dose-escalating design.
Recommended Phase 2 Dose for NAC administered with PBT | From the start date of treatment until 6 months after removal of treatment due to toxicity, termination of study or withdrawal of treatment, whichever came first.
  Determination of the recommended Phase 2 dose (RP2D) will be utilized to evaluate the safety and tolerability of adding NAC to PBT.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Bota, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center